CLINICAL TRIAL: NCT04854122
Title: The Effects of Exercise Training on Central and Peripheral Blood Flow Regulation in Individuals With Down Syndrome
Brief Title: Blood Flow Regulation in Individuals With Down Syndrome - Training Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UNLV_BFDS_TrainingStudy; 4R00HD092606-03 (NIH)
Record Dates: First submitted 2020-08-06; First posted 2021-04-22 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Down Syndrome
Keywords: exercise; blood flow regulation; blood pressure; heart rate
MeSH Terms: conditions — Down Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: This intervention study will be set up as a randomized controlled trial comparing the effects of a 12-weeks exercise program to 12-weeks of non-exercise usual care in participants with Down syndrome.
Masking Description: As this is an exercise intervention, both the study team and the participant will be aware of which group the participant is assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined exercise intervention Down syndrome (Experimental): The exercise intervention will last 12 weeks and will consist of a supervised combined aerobic and resistance training program with a frequency of 3 days/week.In the exercise sessions, the participant will work with the trainer on their strength, balance and aerobic endurance. Each session consists of 10 min of strength exercises (Foundational Exercise), 10 min of Hip Strengthening, 10 min of Vestibular and Balance Exercise, and 20 min of Aerobic Exercise, and starts with a warming up and ends with stretching/cooling down. Each new exercise will be introduced in easy steps and practiced until the participant is comfortable executing it.
  Interventions: Behavioral: Combined exercise intervention
- Usual care Down Syndrome (Sham Comparator): The control condition consists of usual activities.
  Interventions: Behavioral: Usual care / Sham intervention
- Reference group without Down syndrome (No Intervention): This reference group of age- and sex-matched inactive individuals without Down syndrome will undergo the same baseline testing as the other groups but without intervention or post-intervention measures.

INTERVENTIONS:
Behavioral: Combined exercise intervention — The exercise intervention will last 12 weeks and will consist of a supervised combined aerobic and resistance training program with a frequency of 3 days/week. Aerobic exercise will be part of all three sessions, with resistance exercise during two out of three sessions. Training sessions will be supervised by personal trainers to ensure the safe use of the equipment and the correct form when performing each exercise. The first 3 weeks of the intervention will be familiarization with the exercises and the program. After a warm-up, the participant will perform 30 min of aerobic exercise at a heart rate of 65% of the participant's maximum heart rate [43], which increases to 65-85% during weeks 4-12 of the intervention. The resistance exercise part will include all major muscle groups, both upper and lower body.
  Arms: Combined exercise intervention Down syndrome
Behavioral: Usual care / Sham intervention — The control condition consists of usual activities.
  Arms: Usual care Down Syndrome

SUMMARY:
Work capacity is an important predictor of declining health or physical function, and of mortality, and is commonly measured as peak oxygen consumption. Peak oxygen consumption is very low in individuals with Down syndrome, the most prevalent genetic cause of intellectual disability. Previous research suggests individuals with Down syndrome may experience a double disadvantage when they are exercising: they may not be able to increase cardiac output sufficiently and they may not be able to allocate adequate blood flow to the working muscles. The aim of this research proposal is therefore to investigate the responses in central and peripheral blood flow regulation and cardiac autonomic function to exercise training in individuals with DS. Additionally the effects of exercise on gait, balance and attitude towards exercise in individuals with DS are investigated.

DETAILED DESCRIPTION:
Down syndrome (DS) is the most prevalent genetic cause of intellectual disability and occurs in approximately 1 in every 700 births in the US. Individuals with DS are at increased risk for a number of health issues. Work capacity is an important predictor of declining health or physical function, and of mortality, and is commonly measured as peak oxygen consumption. Peak oxygen consumption is very low in individuals with DS, and cannot be explained by physical inactivity, lack of motivation, or lack of understanding of the test. To date, the nature of the limitations in work capacity in DS is unknown, and the proposed research aims to address this knowledge gap.

Work capacity is determined by central and peripheral regulation of blood flow (i.e. cardiac output and maintaining arterial blood pressure vs. supplying exercising muscles with oxygen and nutrients). These factors are governed by the sympathetic and parasympathetic branches of the autonomic nervous system. Central regulation of blood flow is impaired in individuals with DS due to cardiovascular autonomic dysfunction, whereby parasympathetic activity is high and sympathetic control is reduced. This results in lower heart rate, less adequate blood pressure control and attenuated catecholamine levels during exercise. It is unknown to what extent this impaired central control impacts cardiac output, and subsequently work capacity, during exercise in individuals with DS.

Peripheral blood flow regulation is even less studied in individuals with DS. Peripheral regulation involves sympathetically regulated vasoconstriction in non-active muscles and tissues, and local mechanisms regulating vasodilation in working muscles, which facilitates blood flow to working muscle in order to meet metabolic demand. Individuals with DS may partly experience reduced work capacity due to this inability to shunt blood to the working tissue effectively. Our pilot data supports this hypothesis in that individuals with DS are unable to vasoconstrict in response to lower body negative pressure, a known sympathoexcitatory maneuver that produces vasoconstriction in controls without disabilities. Importantly, the impact of their lack of sympathetically mediated vasoconstriction on exercise has not been studied, and neither have the local mechanisms regulating appropriate vasodilation in working muscles.

The aim of this research proposal is therefore to determine the impact of limitations in central and peripheral regulation of blood flow on work capacity in individuals with DS. The aim is to examine the responses to exercise training to better understand the underlying mechanisms and the potential to improve health by using this knowledge in exercise interventions.

Overall Aim: To investigate the responses in central and peripheral blood flow regulation and cardiac autonomic function to exercise training in individuals with DS Aim 1: To determine if exercise training improves peripheral or central regulation of blood flow in individuals with DS. The investigators hypothesize that improvements in work capacity in response to chronic exercise training are primarily due to improvements in peripheral blood flow regulation.

Aim 2: To determine if exercise training improves the cardiovascular autonomic profile in individuals with DS The investigators hypothesize that exercise training will improve the response to clinical cardiovascular autonomic tests in individuals with DS.

Aim 3: To determine if exercise training improves gait, balance and attitude towards exercise in individuals with Down syndrome compared to individuals with Down syndrome in a control group and to individuals without DS.

Individuals with DS may experience a double disadvantage when they are exercising: they may not be able to increase cardiac output sufficiently and they may not be able to allocate adequate blood flow to the working muscles. By revealing the impact of autonomic regulation of blood flow in individuals with DS, the results of this project will identify critical aspects needed to improve clinical practice and design of exercise interventions that optimally improve health and functioning.

General study design Intervention. The exercise intervention will last 12 weeks and will consist of a supervised combined aerobic and resistance training program with a frequency of 3 days/week. Aerobic exercise will be part of all three sessions, with resistance exercise during two out of three sessions. Training sessions will be supervised by two instructors to ensure the safe use of the equipment and the correct form when performing each exercise. The first 3 weeks of the intervention will be familiarization with the exercises and the program. After a warm-up, the participant will perform 30 min of aerobic exercise at a heart rate of 65% of the participant's maximum heart rate [43], which increases to 65-85% during weeks 4-12 of the intervention. The resistance exercise part will include all major muscle groups, both upper and lower body, using multi- and single-joint exercises. The exercise load will be selected to ensure fatigue is reached at 12 repetitions (12-RM). Additionally, if the participants are able to complete 14 repetitions for 2 consecutive sessions using proper technique, the load will be increased by 10% of their 12-RM. The control condition consists of usual care with creative activities that do not involve exercise. Familiarization with the intervention will take place in the first three weeks of the intervention, in which the instructors will support the participants to become familiar with the exercises.

Baseline measures Participants will be tested in a postprandial state (>3 h) on 2 separate days and will refrain from exercise 24 h before each test day. Participants will be also asked to refrain from drinking or eating caffeine and drinking alcohol on testing days. Participants who do not follow the requirements on study days will be asked to come back another day. During the first visit, height, weight and circumferences will be measured. Body composition will be determined with a dual energy X-ray absorptiometry (DEXA) scan, to determine forearm composition and mass. Two-dimensional echocardiography (Hitachi Aloka Alpha 7 system, Tokyo, Japan) will be used to measure aortic root diameter, cardiac output, and stroke volume and end systolic volume at rest. In addition, clinical autonomic function tests (heart rate variability at rest and recovery after exercise, deep breathing, Valsalva maneuver, isometric exercise, active and passive orthostasis) will be evaluated during the first study visit.

Familiarization sessions. Parents/care givers are involved in order to provide a supportive environment for participants and to enhance the parent/caregiver understanding of the research. Prior to study initiation, photographs and video clips of the laboratory and study equipment will be provided to help the participants become comfortable with the laboratory environment and equipment, and the informed consent information is sent to the participants and their parents/care-givers for their review. Familiarization for the participants with Down syndrome will be divided in two parts: they will practice and become accustomed with the treadmill and the equipment for the graded maximal exercise test (first visit), and they will practice and become accustomed with the procedures for the hand grip exercise protocol and the lower body negative pressure chamber (LBNP) (second visit).

Descriptions data collection visits (for both pre and post intervention):

During the first data collections visit, after discussing the study and potential questions, participants (and/or parents/caregivers for the group with Down syndrome) will complete a health history questionnaire and physical activity questionnaire to confirm eligibility. For women of childbearing age, the first visit will include a urine pregnancy test using a test stick. Females will be studied during the first 3-5 days of menses or during the placebo phase if taking oral contraceptives, in order to control for hormonal variation. Eligible participants with Down syndrome and their parent/care-giver will then provide written informed consent, or give verbal assent (for individuals with Down syndrome), and the eligible control participants will provide informed consent themselves. For participants with Down syndrome, the first visit continues with baseline measures and familiarization with the graded maximal exercise test protocol. If necessary, additional familiarization sessions will be scheduled for people with Down syndrome. The second visit, the participant performs the graded maximal exercise test and familiarize the participant with the procedures for the third visit: the hand grip exercise protocol and the LBNP. Gait, balance and foot posture will also be measured. The third visit peripheral blood flow will be assessed during the hand grip exercise protocol without and with the LBNP. For control subjects, the first and second visit are combined. Their second visit is the same as the third visit for individuals with Down syndrome.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* sedentary (defined as being involved in less than 30 minutes of moderately-intense physical activity per day)
* additionally for the participants with Down syndrome:
* diagnosis of Down syndrome trisomy 21 and
* normal thyroid function or stable thyroid function (and medications) for at least 6 mo.

Exclusion Criteria:

* congenital heart disease;
* atherosclerotic or other vascular disease;
* asthma or other pulmonary disease;
* hypertension (defined BP >140/90 mmHg);
* blood pressure below 90/60 mmHg;
* history of pre-syncope or syncope;
* diabetes (defined as Hba1c of >7.5% or use of glucose lowering medication);
* severe obesity (defined as BMI >40);
* medications affecting heart rate, blood pressure or arterial function;
* anti-inflammatory medication including NSAIDS;
* current smoking and
* pregnancy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thessa Hilgenkamp, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
De-identified IPD will be made available to other researchers upon request.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of individuals with Down syndrome occurred through flyers and newsletters spread on campus and in support groups, day programs and organizations for individuals with Down syndrome. All communication, including electronic communication and social media, was only used to spread information about the study. All individuals interested in this study (or their caregivers) were asked to initiate contact with the study team for further information about the study and eligibility screening.
Pre-assignment Details: No significant events occurred between the enrollment and assignment of participants to an arm or group.
Period: Overall Study
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Started | 20 | 20 | 20
Completed | 19 | 19 | 20
Not Completed | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: No deviations from participants assigned to the arms in the participant flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age in years, continuous
  Years | 25.70 (3.92) | 25.55 (4.67) | 23.1 (3.34) | 24.78 (4.13)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex, dichotomous, female, male
  Participants
    Female | 12 | 11 | 16 | 39
    Male | 8 | 9 | 4 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race according to NIH categories
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 3 | 2 | 10 | 15
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 1 | 1 | 1 | 3
    White | 14 | 13 | 3 | 30
    More than one race | 1 | 2 | 2 | 5
    Unknown or Not Reported | 1 | 2 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity (Hispanic/Non-Hispanic)
  Participants
    Hispanic or Latino | 1 | 2 | 5 | 8
    Not Hispanic or Latino | 19 | 18 | 14 | 51
    Unknown or Not Reported | 0 | 0 | 1 | 1
Weight [Mean (Standard Deviation); unit: kg] — Weight in kg
  kg | 75.82 (18.25) | 71.75 (19.02) | 67.13 (15.96) | 71.56 (17.85)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Work Capacity at 13 Weeks
Description: Change in work capacity from baseline to 13 weeks, as measured by peak oxygen uptake in ml/kg/min with a graded exercise test on a treadmill.
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher, additional 2 participants with missing data. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline, plus 2 participants with missing data
Measure: Mean (Standard Deviation); unit: change in ml/kg/min
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 13 | 14 | 0
change in ml/kg/min | -1.20 (6.89) | -0.18 (6.89) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.660, t-test, 2 sided

2. Secondary Outcome: Change From Baseline Brachial Blood Flow at 13 Weeks
Description: Forearm blood flow and vascular conductance was measured in both the exercising and non-exercising arm using high definition ultrasound (Alpha 7, Aloka-Hitachi). The brachial artery was imaged in dual mode allowing for simultaneous determination of artery diameter (B-mode) and flow velocity (Doppler mode). Blood flow was determined from the following formula: Forearm Blood flow = (Mean blood velocity) x (Brachial Cross Sectional Area) x (60) and expressed as ml/min. Change from baseline to 13 weeks was presented.
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline, additionally 5 participants with missing data.
Measure: Mean (Standard Deviation); unit: Change in ml/min
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 15 | 11 | 0
Change in ml/min | 24.66 (77.57) | -15.87 (77.57) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.196, t-test, 2 sided

3. Secondary Outcome: Change From Baseline Muscle Oxygenation at 13 Weeks
Description: Muscle oxygenation was measured with near-infrared spectrography (NIRS), which is a simple, noninvasive method for measuring the presence of oxygen in muscle. It monitored changes in muscle oxygenation and blood flow during submaximal and maximal exercise. During exercise, the extent to which skeletal muscles deoxygenate varies according to the type of muscle, type of exercise and blood flow response. We analyzed the change from baseline to 13 weeks in percentage of oxygenated blood during hand grip exercise at 30% of maximal voluntary contraction (HGE 30%MVC).
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher, plus n=5 with missing data. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline, additionally 8 participants with missing data.
Measure: Mean (Standard Deviation); unit: Change % of oxygenated blood
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 10 | 7 | 0
Change % of oxygenated blood | -5.27 (12.36) | 0.49 (4.03) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.256, t-test, 2 sided

4. Secondary Outcome: Change From Baseline Cardiac Output (Aortic Blood Flow) at 13 Weeks
Description: Change from baseline to 13 weeks in cardiac output will be measured during a graded maximal test protocol. The ascending aortic blood flow will be measured using continuous Doppler echocardiography using a pedoff probe in the suprasternal notch.
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. This was a challenging measurement, and valid data at both pre and post was only obtained for n=2 in the exercise group and n=2 in the control group.
Measure: Mean (Full Range); unit: Change in ml
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 2 | 2 | 0
Change in ml | 4.26 [1.24 to 7.28] | 0.84 [0.57 to 1.12] |

5. Secondary Outcome: Change From Baseline Autonomic Cardiac Function at Rest at 13 Weeks
Description: Change from baseline to 13 weeks in clinical autonomic function test: heart rate variability during rest measured in root mean square of successive differences (RMSSD) in ms.
Time Frame: 13 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Change in ms
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 10 | 7 | 0
Change in ms | -7.40 (18.52) | 3.71 (13.65) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.198, t-test, 2 sided

6. Secondary Outcome: Change From Baseline Autonomic Cardiac Function During Orthostasis at 13 Weeks
Description: Change from baseline to 13 weeks in clinical autonomic function test: heart rate variability during orthostasis in root mean square of successive differences (RMSSD) in ms
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher, plus n=5 with missing data. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline, additionally 9 participants with missing data.
Measure: Mean (Standard Deviation); unit: Change in ms
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 9 | 7 | 0
Change in ms | 20.33 (26.34) | -4.43 (14.47) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.043, t-test, 2 sided

7. Secondary Outcome: Change From Baseline IL-6 at 13 Weeks
Description: Change from baseline to 13 weeks for interleukin-6 IL-6 (venous blood sample)
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher, plus n=3 with missing data. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline, additionally 5 participants with missing data.
Measure: Mean (Standard Deviation); unit: Change in pg/mL
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 12 | 11 | 0
Change in pg/mL | -0.75 (2.30) | 3.28 (9.22) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.174, t-test, 2 sided

8. Secondary Outcome: Change From Baseline HDL at 13 Weeks
Description: Change from Baseline in High-Density Lipoprotein in venous blood sample
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher, additional 3 participants with missing data. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline, plus 3 participants with missing data
Measure: Mean (Standard Deviation); unit: Change in mg/dL
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 12 | 13 | 0
Change in mg/dL | -3.67 (7.46) | -2.31 (10.04) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.707, t-test, 2 sided

9. Secondary Outcome: Change From Baseline Superoxide Dismutase at 13 Weeks
Description: Change from Baseline to 13 weeks in super oxide dismutase (venous blood sample)
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher, additional 1 participant with missing data. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline, plus 1 participant with missing data
Measure: Mean (Standard Deviation); unit: Change in pg/mL
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 14 | 15 | 0
Change in pg/mL | -0.5510 (2.42) | -0.1576 (0.8743) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.571, t-test, 2 sided

10. Secondary Outcome: Change From Baseline Comfortable Walking Speed at 13 Weeks
Description: Change from Baseline to 13 weeks in Comfortable walking speed in cm/sec
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher, additional 4 participants with missing data. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline, plus 6 participants with missing data
Measure: Mean (Standard Deviation); unit: Change in cm/sec
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 12 | 10 | 0
Change in cm/sec | 5.49 (14.98) | 1.27 (18.31) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.559, t-test, 2 sided

11. Secondary Outcome: Change From Baseline Fast Walking Speed at 13 Weeks
Description: Change from Baseline to 13 weeks in Fast Walking Speed in cm/sec
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher, additional 3 participants with missing data. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline, plus 6 participants with missing data
Measure: Mean (Standard Deviation); unit: Change in cm/sec
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 12 | 10 | 0
Change in cm/sec | 6.96 (19.99) | -1.93 (19.52) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.306, t-test, 2 sided

12. Secondary Outcome: Change From Baseline Functional Reach at 13 Weeks
Description: Change from baseline to 13 week in Functional Reach, which is a balance test to investigate how far the participant can reach measured in cm.
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher, additional 3 participants with missing data. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline, plus 1 participant with missing data
Measure: Mean (Standard Deviation); unit: Change in cm
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 12 | 15 | 0
Change in cm | -0.82 (2.26) | 0.17 (2.41) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.287, t-test, 2 sided

13. Secondary Outcome: Change From Baseline Timed Up and Go at 13 Weeks
Description: Timed Up and Go is a dynamic balance test involving getting up from a chair, walk around a mark and sit back down, the time in sec to complete whole sequence is the outcome. Change was measured from baseline to 13 weeks.
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline, plus 1 participants with missing data
Measure: Mean (Standard Deviation); unit: Change in seconds
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 15 | 15 | 0
Change in seconds | -0.59 (1.56) | -0.34 (2.34) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.725, t-test, 2 sided

14. Secondary Outcome: Change From Baseline Standing Balance at 13 Weeks
Description: The Sensory Organization Test of the Bertec Balance System was used to detect balance problems with standing under different conditions. The purpose of the Sensory Organization Test is to systematically evaluate the components of the balance control system, including the vision, vestibular, and somatosensory systems in order to identify possible abnormalities in these systems. The Sensory Organization Test has 6 separate conditions varying in eyes open/closed, fixed or moving visual environment and fixed or moving support surface. This test provides a quantitative evaluation of the person's sway during the 6 conditions, presented as equilibrium score from 0-100 for each condition, with higher scores representing better equilibrium. The composite score is the average equilibrium score of the six conditions.
Time Frame: 13 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change in Composite score
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 13 | 14 | 0
Change in Composite score | 1.11 (6.71) | -3.39 (9.25) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.163, t-test, 2 sided

15. Other Pre Specified Outcome: Change From Baseline C-Reactive Protein at 13 Weeks
Description: Change from Baseline to 13 weeks in C-Reactive Protein (CRP) in pg/mL (venous blood sample)
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher, additional 1 participant with missing data. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline, plus 2 participants with missing data
Measure: Mean (Standard Deviation); unit: Change in pg/mL
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 14 | 14 | 0
Change in pg/mL | -860792 (1614281) | 457370 (953205) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.014, t-test, 2 sided

16. Other Pre Specified Outcome: Change From Baseline Tumor Necrosis Factor - Alpha at 13 Weeks
Description: Change from Baseline to 13 weeks in Tumor Necrosis Factor - alpha (TNF-alpha) in pg/mL (venous blood sample)
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher, additional 2 participants with missing data. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline, plus 3 participants with missing data
Measure: Mean (Standard Deviation); unit: Change in pg/mL
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 13 | 13 | 0
Change in pg/mL | -1.1142 (2.28008) | 1.1892 (2.98976) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.042, t-test, 2 sided

17. Other Pre Specified Outcome: Change From Baseline Glucose at 13 Weeks
Description: Change from Baseline to 13 weeks in Glucose in mg/dL (venous blood sample)
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher, additional 3 participants with missing data. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline, plus 2 participants with missing data
Measure: Mean (Standard Deviation); unit: Change in mg/dL
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 12 | 14 | 0
Change in mg/dL | 1.41 (16.00) | -0.21 (9.36) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.750, t-test, 2 sided

18. Other Pre Specified Outcome: Change From Baseline Leptin at 13 Weeks
Description: Change from Baseline to 13 weeks in Leptin in pg/mL (venous blood sample)
Time Frame: 13 weeks
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Change in pg/mL
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 14 | 14 | 0
Change in pg/mL | -24203 (30074) | -6216 (37238) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.172, t-test, 2 sided

19. Post Hoc Outcome: Change From Baseline 2-Minute-Step Test (2MST) at 13 Weeks
Description: Change from Baseline to 13 weeks in 2-Minute-Step Test in numbers of steps
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline, plus 1 participant with missing data.
Measure: Mean (Standard Deviation); unit: Change in number of steps
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 15 | 15 | 0
Change in number of steps | 25.47 (18.16) | 12.6 (14.09) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.039, t-test, 2 sided

20. Post Hoc Outcome: Change From Baseline Weight at 13 Weeks
Description: Change from Baseline to 13 weeks in Weight in kg
Time Frame: 13 weeks
Population: No post data collection for reference group without Down syndrome. Exercise group DS: 4 participants excluded due to not compliant with exercise group requirements of 20 minutes at 65%HR or higher. Usual care group DS: 3 participant excluded due to >100% increase in physical activity and being classified in the highest IPAQ physical activity category at post data collection compared to lowest category at baseline.
Measure: Mean (Standard Deviation); unit: Change in kg
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 15 | 16 | 0
Change in kg | -0.93 (2.18) | -0.0312 (1.51) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.191, t-test, 2 sided

21. Post Hoc Outcome: Change From Baseline Waist Circumference at 13 Weeks
Description: Change from Baseline to 13 weeks in Waist Circumference in cm
Time Frame: 13 weeks
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Change in cm
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 14 | 14 | 0
Change in cm | -1.43 (3.44) | 1.71 (3.98) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.034, t-test, 2 sided

22. Post Hoc Outcome: Change From Baseline BMI at 13 Weeks
Description: Change from Baseline to 13 weeks in BMI in kg/m2
Time Frame: 13 weeks
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Change in kg/m2
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
Number analyzed (Participants) | 15 | 16 | 0
Change in kg/m2 | -0.38 (1.06) | 0.15 (1.00) |
Statistical Analysis 1: Comparison: Combined Exercise Intervention Down Syndrome vs Usual Care Down Syndrome; Test type: Superiority; p = 0.162, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From baseline data collection until end of post-data collection, up to 3 months.
Arm/Group | Combined Exercise Intervention Down Syndrome | Usual Care Down Syndrome | Reference Group Without Down Syndrome
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT04854122/Prot_SAP_000.pdf
  • Informed Consent Form: Informed Consent Form Reference group no Down Syndrome (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT04854122/ICF_001.pdf
  • Informed Consent Form: Informed Consent Form Down Syndrome (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT04854122/ICF_002.pdf